CLINICAL TRIAL: NCT03795493
Title: Diet Restriction and Exercise-induced Adaptations in Metastatic Breast Cancer
Acronym: DREAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Cancer Society (CCS) (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HREBA.CC-18-0657
Record Dates: First submitted 2018-11-26; First posted 2019-01-07 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Exercise; Nutrition; Caloric Restriction; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Standard chemotherapy treatment and oncology care plus short-term diet and exercise intervention.
  Interventions: Behavioral: Short-term diet and exercise intervention
- Control Group (No Intervention): Standard chemotherapy treatment and oncology care.

INTERVENTIONS:
Behavioral: Short-term diet and exercise intervention — Participants assigned to the intervention group will perform both the diet and acute exercise interventions. The interventions will be applied prior to up to six chemotherapy cycles of a consistent protocol. The total number of treatments of a given protocol received prior to treatment conclusion is dependent on patient condition and oncologic care preferences.
  Arms: Intervention Group

SUMMARY:
Fifty patients with metastatic breast cancer will be randomly assigned to an acute intervention consisting of both aerobic exercise and caloric restriction administered acutely prior to each of six chemotherapy cycles, or to usual care. The aerobic exercise intervention will consist of a single supervised recumbent cycle ergometer session performed concurrent to each chemotherapy infusion. The diet intervention consists of provision of meals freshly prepared in a metabolic kitchen with caloric content equivalent to 50% of measured energy requirements and low carbohydrate content for 48-72 hours prior to each chemotherapy infusion. Tumor outcomes will be assessed via CT scan (tumor size) and MRI (novel marker of tumor regression), while treatment side effects will be assessed by MRI and treatment symptoms and quality of life will be assessed via questionnaire before, during and after up to six chemotherapy cycles of a consistent treatment protocol. Progression-free and overall survival will be tracked for two years after diagnosis.

DETAILED DESCRIPTION:
Despite major advances in recent decades in treatment for early stage breast cancer leading to an 89% 5-year survival rate, metastatic breast cancer is still considered incurable due to resistance to most available treatments. As such, 5-year survival rate for metastatic breast cancer is only 22%. One mechanism for resistance to cancer therapies and promotion of metastasis in solid tumors is that their vascular system is impaired causing diminished delivery of systemic therapy and oxygen. Furthermore, toxicity can be quite high with metastatic regimens, which can limit the dose received. Both diet and exercise have been used to attenuate treatment toxicity, but the promising preclinical evidence showing their potential to enhance chemotherapy efficacy and survival has not been studied in humans. For example, a single bout of aerobic exercise substantially increased tumor blood flow and oxygen delivery, suggesting that chemotherapy delivery to the tumor would be enhanced. Short periods of fasting or caloric restriction also appear to be safe and effective strategies to inhibit tumor growth and enhance chemotherapy efficacy, while also promoting resistance to chemotherapy in healthy cells. Furthermore, combining aerobic exercise and caloric restriction can elicit synergistic effects on outcomes relevant to cancer, including body composition, aerobic fitness, fasting insulin and glucose, insulin-like growth factor, and tumor promoter pathways.

Study Design: With preclinical proof-of-principle and clinical safety and feasibility of each intervention independently established, this study will be a phase II, two-arm, single blind, randomized controlled trial. Fifty patients will be randomly assigned to an acute intervention consisting of both caloric restriction administered acutely prior to and aerobic exercise during each treatment of six chemotherapy cycles, or to usual care.

Approach: Participants will include adults with metastatic breast cancer with measurable metastases that will receive intravenous chemotherapy. The aerobic exercise intervention will consist of a single supervised recumbent cycle ergometer session performed concurrent to each chemotherapy infusion. The diet intervention consists of provision of meals freshly prepared in a metabolic kitchen with caloric content equivalent to 50% of measured energy requirements and low carbohydrate content for 48-72 hours prior to each chemotherapy infusion. The diet period will be reduced from 72 to 48 hours when there are <7 days between infusions (ie weekly protocols) to avoid inducing a sustained caloric deficit leading to weight loss. This acute intervention does not lead to long-term nutritional imbalances. Exercise intensity and meals will be individualized to participant abilities and preferences. All participants, regardless of group assignment, will receive a one-time phone consultation with a registered dietitian and a certified exercise physiologist to enhance recruitment and retention. Tumor outcomes will be assessed via CT scan (tumor size) and MRI (novel marker of tumor regression), while treatment side effects will be assessed by MRI and treatment symptoms and quality of life will be assessed via questionnaire before, during and after up to six chemotherapy cycles of a consistent treatment protocol. Progression-free and overall survival will be tracked for two years after diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage IV or metastatic breast cancer;
* Measurable metastases.
* Age >18
* Starting (or having only received one treatment of) any type of intravenously administered chemotherapy;
* Eastern Cooperative Oncology Group (ECOG) Score < 3
* Oncologist approval to participate
* Able to communicate and read and understand English;
* Willing and able to adhere to the study interventions and assessments;

Exclusion Criteria:

* Limitations to sustained exercise (including bone metastases in the femur neck);
* Clinical evidence of cachexia (oncologist's discretion, study team will use body mass index <18.5kg/m² as a flag to highlight concern to treating oncologist);
* Body mass >109 kg at time of enrollment;
* Diabetes;
* Severe food allergies;
* History of eating disorder (diagnosed or self-reported);
* Strict diet restrictions including vegetarian or vegan;
* Unable to provide informed consent (i.e. cognitive impairment);
* Supplemental oxygen requirement;
* Uncontrolled pleural effusions (oncologists approval if pleural effusions exists and are controlled);
* Bilirubin >30 umol/L;
* Creatinine >120 umol/L;
* Pregnant;
* Contraindications to 3T MRI for research purposes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Tumor size change after 6 cycles (mm) | 0-6 weeks before the first chemotherapy treatment of the first cycle and 1-4 weeks after the last chemotherapy treatment of the last cycle
  Change in tumor size measured by computerized tomography after 6 cycles.

SECONDARY OUTCOMES:
Tumor response to therapy by magnetic resonance imaging (mm²/s) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  Magnetic resonance imaging (MRI) derived water apparent diffusion coefficient within the tumor
Tumor size change after 3 cycles (mm) | 0-6 weeks before the first chemotherapy treatment of the first cycle and 1-3 weeks after the last chemotherapy treatment of the third cycle
  Change in tumor size measured by computerized tomography after 3 cycles.

OTHER OUTCOMES:
Left ventricular ejection fraction (%) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  MRI-derived left ventricular ejection fraction
Left ventricular global longitudinal strain (%) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  MRI-derived left ventricular global longitudinal strain
Left ventricular mass (g/m²) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  MRI-derived left ventricular mass
Liver fat fraction (%) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  Percent of fat in liver derived by PROFIT1 chemical-shift encoded MRI
Liver T1 relaxation time (ms) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  MRI-derived relaxation time from healthy liver
Thigh skeletal muscle T1 relaxation time (ms) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  MRI-derived skeletal muscle T1 relaxation time at mid-thigh
Thigh muscle volume (mL) | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  PROFIT1 chemical-shift encoded MRI of the mid-thigh will be used to assess thigh muscle volume
Thigh skeletal muscle fat fraction % | 0-2 weeks before the first chemotherapy treatment of the first cycle and 2-3 weeks after the last chemotherapy treatment of the last cycle
  Percent of intermuscular fat in thigh muscle derived by PROFIT1 chemical-shift encoded MRI
Patient-reported treatment symptoms | 0-2 weeks before the first chemotherapy treatment of the first cycle, at each chemotherapy treatment, and 2-3 weeks after the last chemotherapy treatment of the last cycle
  Patient-reported treatment symptoms assessed using the Rotterdam Symptom Checklist
Self reported quality of life | 0-2 weeks before the first chemotherapy treatment of the first cycle, at the first chemotherapy treatment of 4th cycle, and 2-3 weeks after the last chemotherapy treatment of the last cycle
  Quality of life assessed using the total score from the Functional Assessment of Cancer Therapy - Fatigue Questionnaire. Scores can range from 0 - 52 where a high score represents a better quality of life.
Fatigue | 0-2 weeks before the first chemotherapy treatment of the first cycle, at the first chemotherapy treatment of 4th cycle, and 2-3 weeks after the last chemotherapy treatment of the last cycle
  Fatigue assessed using the total score from the Functional Assessment of Cancer Therapy - Fatigue Questionnaire. Scores can range from 0 - 52 where a high score represents a lower level of fatigue.
Progression-free survival (months) | Two years after study enrollment
  Progression-free survival time extracted from Cancer Control Alberta's electronic database
Overall survival (months) | Two years after study enrollment
  Overall survival time extracted from Cancer Control Alberta's electronic database

CONTACTS AND LOCATIONS:
Overall Officials: Carla Prado, PhD, Principal Investigator — University of Alberta; Richard Thompson, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kirkham AA, King K, Joy AA, Pelletier AB, Mackey JR, Young K, Zhu X, Meza-Junco J, Basi SK, Hiller JP, Brkin T, Michalowski B, Pituskin E, Paterson DI, Courneya KS, Thompson RB, Prado CM. Rationale and design of the Diet Restriction and Exercise-induced Adaptations in Metastatic breast cancer (DREAM) study: a 2-arm, parallel-group, phase II, randomized control trial of a short-term, calorie-restricted, and ketogenic diet plus exercise during intravenous chemotherapy versus usual care. BMC Cancer. 2021 Oct 10;21(1):1093. doi: 10.1186/s12885-021-08808-2. PMID 34629067